CLINICAL TRIAL: NCT06936072
Title: Temporomandibular Joint Eminence Augmentation Using Titanium Ring Inlay: A New Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinai University (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Moawed Ibrahim Ghoneim, PhD, Associate professor of Oral and Maxillofacial Surgery, Sinai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMS 1-04-024
Record Dates: First submitted 2025-04-05; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: TMJ; Augmentation; TMJ - Oral &Amp;Maxillofacial Surgery
Keywords: TMJ; TMJ augmentation; Augmentation; Oral and Maxillofacial surgery

STUDY DESIGN:
Intervention Model Description: A prospective study was conducted on 100 patients (28 males, 72 females; age range: 25-41 years) with TMJ Temporomandibular joint eminence augmentation. Study was performed after ethical approval from Research Ethics Committee, Faculty of Dentistry, Sinai University OMS 01-04-024.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Titanium Ring Inlay Eminence Augmentation Group (Experimental): Procedure:
  Novel titanium ring inlay eminence augmentation via modified ESS technique
  Inverted L-shaped osteotomy with controlled greenstick fracture
  Precise titanium ring (12-15mm diameter) implantation
  Surgical Protocol:
  * Preauricular approach with subperiosteal dissection
  * Dual osteotomy (transverse mid-eminence + vertical parallel to skull base)
  * Titanium ring inlay placement with anatomical contouring
  * Intraoperative functional assessment
  Postoperative Care:
  * Standardized analgesic protocol
  * Physiotherapy protocol initiation at 2 weeks
  * Gradual return to function protocol
  Follow-up Schedule:
  * Clinical assessments at 5 timepoints (T0-T4)
  * Standardized outcome measurements (VAS, MIO, etc.)
  Key Characteristics:
  Single-arm interventional design
  All participants receive identical surgical protocol
  Standardized outcome assessment methodology
  Blinded evaluators for outcome measures (where applicable)
  Rationale for Single Arm Design:
  First-in-human evaluation of nov
  Interventions: Procedure: Titanium Ring Inlay Eminence Augmentation

INTERVENTIONS:
Procedure: Titanium Ring Inlay Eminence Augmentation — * Preauricular approach with subperiosteal dissection
  * Dual osteotomy (transverse mid-eminence + vertical parallel to skull base)
  * Titanium ring inlay placement with anatomical contouring
  * Intraoperative functional assessment

SUMMARY:
To evaluate the efficacy of titanium ring inlay in ESS technique in Temporomandibular joint eminence augmentation

DETAILED DESCRIPTION:
Background:Temporomandibular joint (TMJ) disorders affect approximately 5-12% of the population, with eminence augmentation being a challenging surgical intervention. Current techniques using autogenous grafts or alloplastic materials present limitations including donor site morbidity, resorption, and implant failure. This study evaluates a novel titanium ring inlay technique for TMJ eminence augmentation, which may offer improved stability, osseointegration, and functional outcomes.

Patients and Methods: A prospective study was conducted on 100 patients (28 males, 72 females; age range: 25-41 years) with TMJ Temporomandibular joint eminence augmentation. Study was performed after ethical approval from Research Ethics Committee, Faculty of Dentistry, Sinai University OMS 01-04-024; . Titanium ring inlay procedure was performed to Temporomandibular joint eminence augmentation. Preoperative and postoperative assessments included pain levels (VAS pain), maximum mouth opening (MMO), Clicking during mouth opening, Headach presence, tinnitus and subjective patient feedback.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed TMJ dysfunction requiring eminence augmentation
* Failed conservative management (≥3 months)
* Adequate bone stock for inlay placement
* Willingness to comply with follow-up protocol

Exclusion Criteria:

* Systemic conditions contraindicating surgery
* Active TMJ infection
* Previous TMJ surgery
* Pregnancy
* Neuromuscular disorders-

Ages: 25 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Functional improvement | Baseline (T0); T1 (1 months postoperative); T2 (3 months postoperative); T3 (6 months postoperative); T4 (12 months postoperative).
  Measuring the Maximal interincisal opening (MIO; mm)

SECONDARY OUTCOMES:
Pain Score | Baseline (T0); T1 (1 months postoperative); T2 (3 months postoperative); T3 (6 months postoperative); T4 (12 months postoperative).
  Measuring the Visual Analogue Scale (VAS), pain score (1-10)
Headache | Baseline (T0); T1 (1 months postoperative); T2 (3 months postoperative); T3 (6 months postoperative); T4 (12 months postoperative).
  Measuring the Headache Assessment Presence Yes/No
Tinnitus | Baseline (T0); T1 (1 months postoperative); T2 (3 months postoperative); T3 (6 months postoperative); T4 (12 months postoperative).
  Tinnitus presence (Y/N)

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Faculty of Medicine, University Hospital, Menoufia University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
A prospective study was conducted on 100 patients (28 males, 72 females; age range: 25-41 years) with TMJ Temporomandibular joint eminence augmentation. Study was performed after ethical approval from Research Ethics Committee.